CLINICAL TRIAL: NCT05860075
Title: A Phase 1 Clinical Study to Evaluate IMM01 Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity in Patients With Refractory or Recurrent Hematologic Malignancy
Brief Title: Exploratory Study of IMM01 for Injection in the Treatment of Refractory or Recurrent Hematologic Malignancy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No expected efficacy was observed in subsequent extended phase.The company decided to initiatively terminate the development of IMM01 as monotherapy and fully promote clinical development of combination therapy.
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM01-I
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open-label, dose-escalation and cohort-expansion phase I clinical study to evaluate the safety and tolerability, pharmacokinetics profile, efficacy and immunogenicity of IMM01 in subjects with relapsed or refractory lymphoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMM01 in subjects with hematologic malignancy (Experimental): The escalation dosing were 3µg/kg, 10µg/kg, 50µg/kg, 150µg/kg, 500µg/kg, 1.0mg/kg, 1.5mg/kg and 2.0mg/kg.
  The extend cohorts were Hodgkin's lymphoma, B-cell lymphoma,NK/T-cell lymphoma,AML,MDS and MM cohorts
  Interventions: Drug: IMM01

INTERVENTIONS:
Drug: IMM01 — IMM01 will be administered once a week for 4 weeks.
  Other Names: IMM01 is a recombinant human signal regulatory protein α (SIRPα) IgG1 fusion protein

SUMMARY:
This is a multi-center, open-label, dose-escalation and cohort-expansion phase I clinical study to evaluate the safety and tolerability, pharmacokinetics profile, efficacy and immunogenicity of IMM01 in subjects with refractory or recurrent hematologic malignancy.

DETAILED DESCRIPTION:
IMM01 is administered via intravenous infusion once week of cycle 1- 12 (4 weeks per cycle).

The accelerated titration method and the traditional "3+3" method will be adopted to determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) in dose-escalation phase.

Once the RP2D is determined, will explore for Classic Hodgkin's lymphoma, B-cell lymphoma,NK/T-cell lymphoma, AML, MDS and MM cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. They are voluntary to sign an informed consent form, agree to follow and have the ability to complete all trial procedures with knowledge of the study;
2. Male or female, aged ≥18 and ≤ 75 years;
3. Patients with refractory or recurrent lymphoma diagnosed according to the 2016 WHO classification criteria; the relapsed, refractory lymphoma is defined as follows: Relapse is considered to occur when a new lesion appears at the primary site or elsewhere when response has been achieved with at least one current standard or commonly used regimen;

   Lymphoma is considered refractory if one of the following conditions is met:

   Less than 50% tumor shrinkage or disease progression occurs after ≥4 cycles of treatment with current standard or commonly used regimens; Patients who have achieved partial or complete response by current standard or commonly used regimens and relapsed within six months after termination of treatment;
4. There is at least one measurable or evaluable tumor lesion (preferentially enrolled the measurable lesions), measurable lesions: lymph nodes with longest diameterof ≥15 mm, metastatic lesions (≥10 mm) at other sites; lesions previously treated with local therapy such as radiotherapy are considered measurable lesions if disease progression has been demonstrated;
5. Patients with a performance status score of 0~2 according to the Eastern Cooperative Oncology Group (ECOG) scale;
6. Expected life expectancy of at least 3 months;
7. If prior anti-tumor therapy has been received , the interval to the first dose in this study should meet the following conditions: Those who have used chemotherapy drugs previously need to discontinue for more than 4 weeks.Those with a history of surgery, targeted therapy (including anti CD20 monoclonal antibodies such as rituximab; CD30 monoclonal antibodies such as Brentuximab Vedotin), therapy with anti tumor indications, and palliative radiotherapy should discontinue the treatment for more than 4 weeks;Those with prior CAR-T cell therapy or PD-1/PD-L1 monoclonal antibody therapy need to discontinue for at least 8 weeks;And they have recovered from toxic reactions to previous treatment to grade ≤ 1 identified by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (NCI CTCAE v5.0) (except for residual alopecia).
8. Suitable organs and hematopoietic functions are available. Absolute neutrophil count (ANC) ≥1.0×109/L (no use of short-acting leucopenia drugs within 1 week or no use of long-acting leucopenia drugs within 3 weeks). Patients have not received platelet transfusion within 1 week; platelets

   ≥75×109/L (without bone marrow infiltration)/ ≥50.0×109/L (with bone marrow infiltration).

   Patients have not received red blood cell transfusion within 2 weeks; hemoglobin ≥90 g/L (without bone marrow infiltration)/ ≥70 g/L (with bone marrow infiltration).

   Serum creatinine ≤ 1.5 times the upper limit of normal (ULN). AST and ALT ≤ 2.0 times ULN; Serum total bilirubin (TBIL) ≤ 2 times ULN; International normalized ratio (INR) ≤ 2 times ULN, or activated partial thromboplastin time (APPT) ≤ 1.5 times ULN;
9. Male subjects and female subjects of childbearing age should agree to take effective contraceptive measures from the time they sign the informed consent until 6 months after the last dos

Exclusion Criteria:

1. Patients with any of the following cannot be enrolled: previous allogeneic hematopoietic stem cell transplantation and other organ transplantation; a history of autologous hematopoietic stem cell transplantation for not more than six months.
2. Patients have participated in clinical trials of other drugs or medical devices within 4 weeks prior to the first dose of this study;
3. Presence of central nervous system metastatic lesion;
4. Patients with previous or current other malignancies (except cured stage IB or lower grade cervical cancer, non-invasive basal cell or squamous cell skin cancer; except other malignancies that have achieved complete response (CR) for >5 years and have not been treated with antineoplastic therapy for 5 years);
5. Subjects with active autoimmune disease, or a history of autoimmune disease with a risk of relapse (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc., see Appendix 6), or patients at high risk (e.g., those requiring immunosuppressive therapy after undergoing organ transplantation).

   However, subjects with the following diseases are allowed to enroll :

   Those with autoimmune hypothyroidism who require hormone replacement therapy only; Those with skin conditions (such as eczema, rash covering less than 10% of the body's surface) that do not require systemic treatment;
6. Patients who have undergone major surgery within 28 d prior to enrollment or who are expected to have major surgery during this study period including the 21 d screening period.
7. Subjects requiring systemic corticosteroids (at a dose equivalent to >10 mg prednisone/d) or other immunosuppressive drugs within 14 d prior to enrollment or during the study period; the the patients meet the following conditions are allowed for enrollment: Subjects are allowed to use topical or inhaled glucocorticoids; Short-term (≤7 days) use of glucocorticoids for the prevention or treatment of non-autoimmune allergic diseases is allowed;
8. Patients with a history of arterial thrombosis or deep vein thrombosis within 6 months prior to enrollment or with evidence or history of bleeding tendency within 2 months prior to enrollment, regardless of severity; partial prothrombin time (APTT) or prothrombin time (PT) > 1.2 × ULN; oral warfarin with an international normalized ratio (INR) > 1.2 × ULN
9. Patients with acute lung disease, interstitial lung disease or pneumonia (except for local interstitial pneumonia induced by radiotherapy), pulmonary fibrosis, acute lung disease, etc.;
10. Systemic diseases that have not been stably controlled after treatment, such as diabetes, severe organic cardiovascular disease, cardiac insufficiency, hypertension, heart block of degree II or higher, myocardial infarction within 6 months and cerebral infarction within 6 months, etc;
11. Patients with positive HIV test;
12. Patients with active tuberculosis disease at screening;
13. Patients with HBsAg (+); with HBsAg (-) but HBV-DNA quantification exceeding the upper limit of the normal; Patients with HCV-Ab (+); with HCV-Ab (-) but HCV-RNA quantification exceeding the upper limit of the normal;
14. Patients with serious infections within 4 weeks prior to the first dose, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
15. Patients with uncontrolled active infectious lesions requiring oral or intravenous antibiotic therapy;
16. Subjects with a history of severe allergy or those who are known to have had severe allergic reactions to large molecular protein preparation/monoclonal antibodies, and any of the components of the investigational drug (greater than grade 3 according to NCI-CTCAE v5.0 classification);
17. Patients with a history of alcohol, drug or substance abuse within the last 1 year;
18. Patients with a clear previous history of neurological or psychiatric disorders with poor compliance, such as epilepsy, dementia;
19. Pregnant and lactating women;
20. Subjects with other conditions not suitable for participating in the study at the investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | 48 weeks of treatment
  Incidence and characteristics of adverse events (AEs), serious adverse events (SAEs)
Dose-limiting toxicities (DLTs) | Evaluated during the first treamtment cycle of 28 days
  Incidence and characteristics of dose-limiting toxicities (DLTs)
Maximum Tolerated Dose（MTD ） | 48 weeks of treatment
  MTD is the highest dose in patients with DLT incidence <30%.

SECONDARY OUTCOMES:
Anti-drug antibody (ADA) | 48 weeks of treatment
  To evaluate the immunogenicity of IMM01 in patients with refractory or recurrent hematologic malignancy
Overall Rate Response (ORR) | When the last subject enrolled completes approximately 48 weeks of treatment
  ORR is defined as the proportion of participants who have a partial response (PR) or critical response (CR)
Disease Control Rate (DCR) | From start of treatment to the last subject enrolled completes approximately 48 weeks of treatment]
  DCR is defined as the proportion of participants who have a critical response (CR), partial response (PR) or disease stable (SD)
Duration of Response (DOR) | From start of treatment to the last subject enrolled completes approximately 48 weeks of treatment
  DOR is defined as time from date of initial documentation of a response (PR or CR) to date of first documented evidence of progressive disease (PD)
Progression-free survival (PFS) | From start of treatment to treatment termination visit, up to 48 weeks
  Defined as the duration from the start of treatment until tumor progression or death of any cause
Maximum Plasma Concentration (Cmax) | 48 weeks of treatment
  Maximum Plasma Concentration observed in patients with IMM01 dosed
time to maximum concentration (Tmax) | 48 weeks of treatment
  time to maximum concentration observed in patients with IMM01 dosed

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College,, Tianjin, Tianjin Municipality, China